CLINICAL TRIAL: NCT05380284
Title: Evaluation of Senior Driving Simulation Training on Executive Function, Cognitive Promotion and EEG in Subjective Cognitive Decline and Mild Cognitive Impairment
Brief Title: Senior Driving Simulation Training for Subjective Cognitive Decline and Mild Cognitive Impairment
Acronym: SDST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Huie-Ling Chiu, Assistant professor, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: N202002083
Record Dates: First submitted 2022-04-30; First posted 2022-05-18 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: MCI; Subjective Cognitive Decline; Healthy Aging
Keywords: driving simulation; executive function; brain wave

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Senior Driving Simulation Training
  Interventions: Other: Senior Driving Simulation Training
- Control Group (Other): Ｗaiting-list
  Interventions: Other: Waiting list control

INTERVENTIONS:
Other: Senior Driving Simulation Training — The experimental group (Senior Driving Simulation Training: 30-mins training session two times per week for 5 weeks, with a total of 10 sessions) .
  Arms: Experimental Group
Other: Waiting list control — The control group is waiting list control. They will also receive the (Senior Driving Simulation Training) after all research is done.
  Arms: Control Group

SUMMARY:
This study aims to establish the Senior Driving Simulation Training (SDST) for Subjective Cognitive Decline (SCD) and Mild Cognitive Impairment (MCI), and explore the effectiveness of Senior Driving Simulation Training (SDST) on the executive function, cognitive function and EEG.

DETAILED DESCRIPTION:
Driving behavior is a high cognitively demanding task, and whether the Subjective Cognitive Decline (SCD) and Mild Cognitive Impairment (MCI) can continue to drive is an important issue. This study will develop the Taiwan version of innovative, immediate feedback and environmentally safe Senior Driving Simulation Training (SDST). This study aims to establish the Senior Driving Simulation Training (SDST) for Subjective Cognitive Decline (SCD) and Mild Cognitive Impairment (MCI), and explore the effectiveness of Senior Driving Simulation Training (SDST) on the executive function, cognitive function and EEG. The investigators intend to conduct a single-blind randomized controlled trial using a two-arm parallel-group design. Participants will be randomized by the permuted block randomization, block size of 4, into an experimental group (Senior Driving Simulation Training: 30-mins training session two times per week for 5 weeks, with a total of 10 sessions) or a control group (Waiting list). The investigators plan to blind the therapists and outcome assessors to maintain the blinding methods' quality. The primary outcome indicators are mental set-shifting, working memory, and inhibition. The secondary outcome indicators are cognitive function and EEG. The investigators also evaluate visual awareness and simulator sickness. The short-term (immediate post-test) and the long-term (3, 6, and 12 months) effectiveness of the intervention on individual outcome measures will be analyzed by the generalized estimating equation. The investigators also plan to use the secondary data analysis methods to investigate the relationship between objective indicators of a driving simulator, executive function, cognitive function, EEG, visual awareness, and simulator sickness. Furthermore, the investigators will analyze the trend of EEG while the participants conducting the training, and complete the psychometric properties of the Chinese version of the Cognitive Change Index (C-CCI). This will be the first senior driving simulation training (SDST) for Subjective Cognitive Decline (SCD) and Mild Cognitive Impairment (MCI) in Taiwan. Results of the current study will provide valuable information on driving safety decisions and apply to promote the advanced driving policies.

ELIGIBILITY:
Inclusion Criteria:

* Subjective cognitive decline( AD-8 scale ≥1 point).
* Mild cognitive impairment (AD-8 scale ≥ 2 points), and MMSE> 24 points, can maintain personal daily activity function.
* Can communicate in Chinese or Taiwanese.
* At least 60 years of age.
* Those with a car driving license.
* No physical impairment.
* In addition to the above conditions, participants must be voluntary and signed informed consent.

Exclusion Criteria:

* Dementia, diagnosed by a physician and in compliance with ICD-10.
* Significant mental illness or communication impairment.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-06-28 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-05-28 (Actual)

PRIMARY OUTCOMES:
Mental set shifting, measured by Wisconsin Card Sorting Test | immediate post-test
  Mental set shifting is one of the sub-categories of executive function
Change from Baseline Mental set shifting, measured by Wisconsin Card Sorting Test at 3 months | 3 months follow-up
  Mental set shifting is one of the sub-categories of executive function
Working memory, measured by Digit span test | immediate post-test
  Working memory is one of the sub-categories of executive function
Change from Baseline Working memory, measured by Digit span test at 3 months | 3 months follow-up
  Working memory is one of the sub-categories of executive function
Inhibition, measured by the Stroop Color and Word Test | immediate post-test
  Inhibition is one of the sub-categories of executive function
Change from Baseline Inhibition, measured by the Stroop Color and Word Test at 3 months | 3 months follow-up
  Inhibition is one of the sub-categories of executive function

SECONDARY OUTCOMES:
Cognitive function measured by Montreal Cognitive Assessment | immediate post-test
  Cognitive function measured by Montreal Cognitive Assessment
Cognitive function measured by Cognitive Change Index(C-CCI) | immediate post-test
  Cognitive function measured by Cognitive Change Index(C-CCI)
Change from Baseline cognitive function by Montreal Cognitive Assessment at 3 months | 3 months follow-up
  Change from Baseline cognitive function by Montreal Cognitive Assessment at 3 months
Change from Baseline cognitive function by Cognitive Change Index(C-CCI)at 3 months | 3 months follow-up
  Change from Baseline cognitive function by Cognitive Change Index(C-CCI)at 3 months
EEG | immediate post-test
  EEG power in delta, theta, alpha, and beta band
Change from Baseline EEG at 3 months | 3 months follow-up
  EEG power in delta, theta, alpha, and beta band
Visual awareness measured by CANTAB | immediate post-test
  Visual awareness measured by CANTAB
Visual awareness measured by trail making test | immediate post-test
  Visual awareness measured by trail making test
Change from Baseline visual awareness by CANTAB at 3 months | 3 months follow-up
  Visual awareness measured by CANTAB
Change from Baseline visual awareness by trail making test at 3 months | 3 months follow-up
  Change from Baseline visual awareness by trail making test at 3 months
simulator sickness | immediate post-test
  Simulator Sickness Questionnaire (SSQ). The 16-item SSQ will be used to assess participants' sickness levels. This is the 4-point Likert scale (0 - "None" to 3 - "Severe"), and the higher total score reflects more severe sickness.
Usability | immediate post-test
  The System Usability Scale (SUS) will be used to access the usability, this scale consists of 10 items, and the higher total score reflects better usability.
Acceptance | immediate post-test
  The Technology Acceptance for Older Adults Scale will be used to access the acceptance, this scale consists of 17 items, and the higher total score reflects better acceptance.

CONTACTS AND LOCATIONS:
Overall Officials: Huei-Ling Chiu, Principal Investigator — Taipei Medical University
Locations (1):
- Taipei Medical University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No